CLINICAL TRIAL: NCT06909786
Title: Effect of Intraoperative Implementation of the Hypotension Prediction Index (HPI) Guided Management Strategy on Incidents of Intraoperative Hypotension Among Frail Patients Undergoing Major Abdominal Surgery
Brief Title: Hypotension Prediction Index and Intraoperative Hypotension Incidence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Guan Zheng, associate professor, First Affiliated Hospital Xi'an Jiaotong University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XJTU1AF2024LSYY-152
Record Dates: First submitted 2025-03-23; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Intraoperative Hypotension
Keywords: intraoperative hypotension; hypotension prediction index; frail patient; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard arterial line group (Sham Comparator): BP, ECG and SpO2 were monitored after entering the operating room, peripheral venous access was established, radial artery puncture catheterization under local anesthesia and connected to TruWave DPT and run data via HemoSphere machine (Edwards Lifesciences). The target of intraoperative blood pressure was to maintain MAP > 65mmHg. Timing of treatment and choice of treatment is then left to the discretion of the attending physician.
  Interventions: Other: standard arterial line
- HPI guided hemodynamic management group (Experimental): BP, ECG and SpO2 were monitored after entering the operating room, peripheral venous access was established, radial artery puncture catheterization under local anesthesia and connected to the HPI (Edwards Lifesciences).
  The treating anesthetist is trained to understand Acumen IQ parameters and the meaning of HPI, MAP, CI, SVI, SVR, SVV, Eadyn, dP/dtmax. The treating anesthetist is provided with guidance by means of a flowchart suggesting when to treat and how to treat hypotension. The hemodynamic management is performed according to the HPI guided algorithm.
  Interventions: Procedure: HPI guided hemodynamic management

INTERVENTIONS:
Procedure: HPI guided hemodynamic management — BP, ECG and SpO2 were monitored after entering the operating room, peripheral venous access was established, radial artery puncture catheterization under local anesthesia and connected to the HPI (Edwards Lifesciences).
  The treating anesthetist is trained to understand Acumen IQ parameters and the meaning of HPI, MAP, CI, SVI, SVR, SVV, Eadyn, dP/dtmax. The treating anesthetist is provided with guidance by means of a flowchart suggesting when to treat and how to treat hypotension. The hemodynamic management is performed according to the HPI guided algorithm.
  Arms: HPI guided hemodynamic management group
Other: standard arterial line — BP, ECG and SpO2 were monitored after entering the operating room, peripheral venous access was established, radial artery puncture catheterization under local anesthesia and connected to TruWave DPT and run data via HemoSphere machine (Edwards Lifesciences). The target of intraoperative blood pressure was to maintain MAP > 65mmHg. Timing of treatment and choice of treatment is then left to the discretion of the attending physician.
  Arms: standard arterial line group

SUMMARY:
This study aim to implement intraoperative hemodynamic monitoring and management guided with HPI algorithm in frail patients undergoing elective abdominal surgery. Investigators hypothesize that the use of this algorithm will alter treatment of hypotension and reduces the amount of hypotension as measured by the time weighted average (TWA) during non-cardiac surgery and to anticipate a reduction of postoperative AKI incidents, to explore the clinical benefits of impact of Acumen guided algorithm hemodynamic management in postoperative intestinal function recovery, and postoperative cardiac complications.

DETAILED DESCRIPTION:
Intraoperative hypotension (IOH) is common, a study involved 34,045 surgical patients in elective, emergency, and intensive care unit (ICU) found that the incidence of hypotension (defined as systolic blood pressure below 80mmHg) greater than 5 minutes and 10 minutes was 25.7% and 14.6%, respectively. In another large sample size study of 22,109 patients with ASA grade 3 to 4 undergoing surgery with duration of ≥180 minutes found that 88% of patients experienced at least one episode of intraoperative hypotension, defined as a fall in mean arterial pressure (MAP) below 65 mmHg lasting at least 1 min. A multicenter retrospective cohort study from the U.S. electronic health record database conducted between 2008 and 2017 and including 368222 noncardiac surgeries reported that the incidence of MAP ≤65 mmHg during surgery was 19.3%.

IOH was significantly associated with postoperative complications and poor outcomes. Meta-analysis suggests that IOH increases the incidence of acute kidney injury, myocardial injury, and 30-day mortality after noncardiac surgery. Intraoperative MAP below 70 mmHg is an independent risk factor for increased mortality at 30 days postoperatively, while intraoperative MAP below 65 mmHg is an independent risk factor for myocardial injury after noncardiac surgery. Studies of non-cardiac, non-obstetric surgery have found that intraoperative MAP events below 55 mmHg is associated with persistent renal impairment up to 90 days postoperatively. In addition, intraoperative MAP reductions of more than 30% are associated with postoperative ischemic stroke.

China is experiencing an aging population, the number of elderly patients receiving surgical anesthesia is increasing year by year. Based on the 5-items frailty assessment scale shown that old age is closely related to the development of frailty. The prevalence of frailty among patients over 65-year-old was 7%, and 26% in patients with age over 85 years. Frailty refers to a state in which the functions of multiple systems are cumulatively reduced, leading to a decline in the body's reserve capacity and resistance. Frail patients have decreased organ reserve function, decreased response ability to surgical stress, reduced cardiac stroke volume, impaired cardiac autonomic nervous system function, and decreased albumin levels, resulting in increased blood concentration of anesthetic drugs, at risk for persistent hypotension and severe postoperative complications. In addition, the occurrence of intraoperative hypotension may further aggravate organ dysfunction on the impaired functionality of ischemia-sensitive organs such as the kidneys. The postoperative complications in frail patients undergoing abdominal surgery is as high as 45.5-57.1%. Therefore, it is important to strengthen intraoperative blood pressure management and prevent hypotensive events in frail patients.

IOH is preventable and may potential to improvement in postoperative outcomes. Futier et al highlighted management targeting an individualized systolic blood pressure, compared with standard management, reduced the risk of postoperative organ dysfunction 30 days after surgery. Current treatment of intraoperative hypotensive episodes is not proactive and rather occurs with some delay. For elderly frail populations undergoing major surgery, there is need for a novel method to prevent hypotension.

Edwards Lifesciences has developed an algorithm that by applying machine learning methods analyzing continuously invasively measured arterial waveforms with the Acumen lQ is able to predict hypotension, defined as a mean arterial pressure (MAP) below 65 mmHg lasting for at least 1 min. The Hypotension Prediction Index (HPI) ranges from 0 to 100, and higher values reflect a higher likelihood of hypotension and shorter intervals between periods of hypotension. In major abdominal surgery, HPI demonstrated a sensitivity of 85.8%, 81.7%, and 80.6% respectively to predict a hypotensive event at 5, 10, and 15 minutes before a hypotensive event. The HPI enable the treating anesthetist to proactive treat the predicted hypotension. Various studies have shown that HPI ability in reducing TWA-MAP < 65mmHg and significantly reduction in the incidence of IOH in major noncardiac surgery such as abdominal surgery, gastrointestinal surgery, spinal surgery, in elderly populations undergoing orthopedics surgery.

This study aim to implement intraoperative hemodynamic monitoring and management guided with HPI algorithm in frail patients undergoing elective abdominal surgery. Investigators hypothesize that the use of this algorithm will alter treatment of hypotension and reduces the amount of hypotension as measured by the time weighted average (TWA) during non-cardiac surgery and to anticipate a reduction of postoperative AKI incidents, to explore the clinical benefits of impact of Acumen guided algorithm hemodynamic management in postoperative intestinal function recovery, and postoperative cardiac complications.

ELIGIBILITY:
Inclusion Criteria:

* Age> 60 years old
* Frail score > 2
* ASA≥2
* Planned to receive general anesthesia
* Elective laparoscopic or laparotomy major abdominal surgery with an expected duration of > 180 minutes
* Planned to receive an arterial line monitoring intraoperatively
* Being able to give written informed consent prior to surgery

Exclusion Criteria:

* Severe cardiac arrhythmia including atrial fibrillation
* Severe aortic stenosis
* Uncontrolled Hypertension (sitting systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥100 mmHg during screening)
* Significant hypotension before surgery defined as a MAP <65mmHg
* Chronic kidney disease with glomerular filtration rate <30 ml/min/1.73 m2 or requiring renal-replacement therapy for end-stage renal disease
* Organ transplant surgery, surgery involving the kidney, liver surgery requiring hilar blockage, surgery requiring controlled hypotension or controlled low central venous pressure

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of intraoperative hypotension | From anesthesia to end of operation, assessed up to 8 hours.
  Definition of intraoperative hypotension: MAP< 65mmHg lasting for> 1 minute. The occurrence of intraoperative hypotension: number of hypotension events, area under the hypotension curve, time-weighted average hypotension, total cumulative time of hypotension, ratio of cumulative total time of hypotension to length of operation

SECONDARY OUTCOMES:
Incidents of AKI | From end of operation to 48 hours after operation, up to 48 hours.
  Definition of AKI according to KDIGO (Kidney Disease Improving Global Outcomes) criteria: elevated serum creatinine more than 0.3 mg/dl within 48 hours or more than 150% of basal value within 7 days, or urine output < 0.5 ml/kg/hour for more than 6 hours. The stages of AKI will not be divided.
Intestinal peristalsis recovery time | From end of operation to first bowel movement, assessed up to 48 hours.
  Auscultation every 4 hours after surgery, and the appearance of ≥4 bowel sounds per minute is considered to be intestinal peristalsis recovery.
Intestinal function recovery time | From end of operation to first passage of flatus, assessed up to 48 hours.
  Time from end of operation to first passage of flatus
Incidence of myocardiac injury | From end of operation to 7 days after operation, up to 7 days.
  Presence of ECG changes (bundle branch block, premature beats, or T-wave changes) or cardiographic enlargement or decreased cardiac function, elevated cTn/T >14 pg/ml and/or CK/MB elevated >8.8 ng/ml.
Incidence of congestive heart failure | From end of operation to 7 days after operation, up to 7 days.
  Pulmonary edema with clinical or radiographic evidence, requiring diuretic or vasodilator therapy, oxygen saturation less than 93% with or without mechanical ventilation.
Incidence of acute myocardial infarction | From end of operation to 7 days after operation, up to 7 days.
  Elevated troponin with at least one of the following: symptoms of myocardial ischemia, new-onset ECG changes (Q-wave formation, left bundle branch block), local ventricular wall motion abnormalities.

OTHER OUTCOMES:
Mechanical ventilation support time | From anesthesia induction to anesthesia recovery, assessed up to 24 hours.
  The duration participants underwent mechanical ventilation.
PACU time | From admitted in PACU to discharged from PACU, assessed up to 24 hours.
  The duration participants admitted in the PACU.
ICU time | From admitted in ICU to discharged from ICU, assessed up to 3 days.
  The duration participants admitted in the ICU
Hospitalization time | From admission to discharge, assessed up to 15 days.
  The duration participants in hospitalization.
Total hospitalization cost | From admission to discharge, assessed up to 15 days.
  Total expenses during hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No